CLINICAL TRIAL: NCT04848480
Title: Efficacy and Safety of Once Weekly Insulin Icodec Compared to Once Daily Insulin Degludec 100 Units/mL, Both in Combination With Insulin Aspart, in Adults With Type 1 Diabetes. A 26-week, Randomised, Multicentre, Open-label, Active-controlled, Parallel Group, Two Armed, Treat-to-target Trial Investigating the Effect on Glycaemic Control and Safety of Treatment With Once Weekly Insulin Icodec Compared to Once Daily Insulin Degludec, Both in Combination With Insulin Aspart in Adults With Type 1 Diabetes, With a 26-week Extension Investigating Long Term Safety
Brief Title: A Research Study to Compare a New Weekly Insulin, Insulin Icodec, and an Available Daily Insulin, Insulin Degludec, Both in Combination With Mealtime Insulin in People With Type 1 Diabetes (ONWARDS 6)
Acronym: ONWARDS 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4625; U1111-1251-7315 (Other: World Health Organization (WHO)); 2020-002374-27 (EudraCT Number)
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec; insulin degludec; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec + insulin aspart (Experimental): insulin icodec once a week in combination with 2-4 times daily injections of insulin aspart at meal times.
  Interventions: Drug: insulin icodec; Drug: insulin aspart
- Insulin degludec + insulin aspart (Active Comparator): insulin degludec once a day in combination with 2-4 times daily injections of insulin aspart at meal times.
  Interventions: Drug: insulin degludec; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin icodec — insulin icodec 700 units/mL, subcutaneously (under the skin), solution for injection once weekly
  Arms: Insulin icodec + insulin aspart
Drug: insulin degludec — insulin degludec 100 units/mL, subcutaneously (under the skin), solution for injection once daily
  Arms: Insulin degludec + insulin aspart
Drug: insulin aspart — insulin aspart 100 units/mL, subcutaneously (under the skin), solution for injection daily

SUMMARY:
This study compares insulin icodec (a new insulin) to insulin degludec (an insulin already available on the market) in people with type 1 diabetes.

The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin degludec taken daily.

Participants will either get insulin icodec that participants will have to inject once a week on the same day of the week, or insulin degludec that participants will have to inject once a day at the same time every day. Which treatment participants get is decided at random. Participants will also get a mealtime insulin.

The insulin is injected with a needle in a skin fold in the thigh, upper arm or stomach.

The study will last for about 1 year and 2 months. Participants will have 28 clinic visits and 28 phone calls with the study doctor. At 11 clinic visits participants will have blood samples taken.

At 6 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Participants will be asked to wear a sensor that measures your blood sugar all the time. Participants will be asked to wear it for a total of 57 weeks (around 1 year).

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged greater than or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 1 diabetes mellitus greater than or equal to 1 year prior to the day of screening.
* Treated with multiple daily insulin injections (basal and bolus insulin analogue regimes) greater than or equal to 1 year prior to the day of screening.
* HbA1c below10% at screening visit based on analysis from central laboratory.

Exclusion Criteria:

* Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days prior to the day of screening.
* Chronic heart failure classified as New York Heart Association (NYHA) Class IV at screening.
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (1452), Study Director — Novo Nordisk A/S
Locations (129):
- United States (41):
  - John Muir Physicians Network, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Valley Research, Fresno, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Diabetes & Endocrine Associates, La Mesa, California
  - Mills-Peninsula Hlth Services, San Mateo, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Northeast Research Institute, Fleming Island, Florida
  - Center For Diabetes & Endo Care, Fort Lauderdale, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - Endo Res Solutions Inc, Roswell, Georgia
  - Northwestern University_Chicago, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Cotton-O'Neil Diab & Endo Ctr, Topeka, Kansas
  - Endo and Metab Consultants, Rockville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - MassResearch, LLC, Waltham, Massachusetts
  - Minn Center For Obesity Met & Endocrinology, Eagan, Minnesota
  - International Diabetes Center, Minneapolis, Minnesota
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - Mercy Research, Springfield, Missouri
  - Methodist Physicians Clin, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern NH Diabetes and Endo_Nashua, Nashua, New Hampshire
  - John J Shelmet, MD, Lawrenceville, New Jersey
  - AMC Community Endocrinology, Albany, New York
  - Accellacare, Wilmington, North Carolina
  - Prisma Health-Upstate, Greenville, South Carolina
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Rainier Clin Res Ctr Inc, Renton, Washington
- Austria (6):
  - Univ.-Klinik für Innere Medizin, Graz
  - Univ.-Klinik für Innere Medizin I, Innsbruck
  - Fließer-Görzer [Ordination], Saint Stefan
  - Klinik Landstraße, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Hietzing, Vienna
- Canada (10):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - LMC Clinical Res Thornhill, Concord, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Centricity Research LMC, Toronto, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - IRCM, Montreal, Quebec
  - Centre de recherché du CHUS, Sherbrooke, Quebec
  - CHU de Quebec-Universite Laval, Québec
- Germany (10):
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - InnoDiab Forschung GmbH, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - Diabetologische Gemeinschaftspraxis Dr. Staudenmeyer und Dr. Schiwietz, Lingen
  - Die Praxis am Ludwigsplatz, Ludwigshafen
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - RED-Institut für medizinische Studien und Fortbildung GmbH, Oldenburg I. Holst
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
- India (8):
  - Diacare diabetes Hormonal Clinic, Ahmedabad, Gujarat
  - Calicut Medical College, Kozhikode, Kerala
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Fortis Heart Institute and Multispeciality Hospital, Mohali, Punjab
  - Care Hospital, Hyderabad
  - Lady Hardinge Medical College, New Delhi
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram
- Italy (7):
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia, Umbria
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - Azienda Ospedaliero Universitaria Careggi MASTER, Florence
  - Osp. San Raffaele Diabetes Research Institute, Dibit 1, Milan
  - Policlinico Umberto I Clinica Medica DH Diabetologia, Roma
  - Master Centre for Italy, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di scienze Mediche e Chirurgiche, Rome
- Japan (7):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Manda Memorial Hospital_Internal Medicine, Sapporo-shi, Hokkaido, Hokkaido, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - The Institute of Medical Science, Asahi Life Foundation_Internal Medicine, Chuo-ku, Tokyo
  - H.E.C Science Clinic, Kanagawa
  - Yuri Ono Clinic, Sapporo-shi, Hokkaido
  - Tokyo Women's Medical University_Metabolism and Diabetology, Tokyo
- Netherlands (7):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Maxima Medisch Centrum, Eindhoven
  - Bethesda Diabetes Research Center en Bethesda ziekenhuis, Hoogeveen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Ikazia Ziekenhuis, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Russia (14):
  - Volosevich First City Clinical Hospital, Arkhangelsk
  - LLC "Clinic of new technologies in Medicine", Dzerzhinskiy
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Endocrinological Dispensary of Department of healthcare ser., Moscow
  - Endocrinology Dpt,Post-Graduate Medical Education Faculty, Moscow
  - SPb SBHI "Snegirev Maternity Hospital No. 6", Saint Petersburg
  - City Consultative & Diagnostic Centre #1, Saint Petersburg
  - SPb SBHI City Multifield Hospital #2, Saint Petersburg
  - SPb SBHI City polyclinic #117, Saint Petersburg
  - LLC "Endocrinolog", Samara
  - SHI Saratov City Clinical Hospital #9, Saratov
  - Saratov regional clinical hospital, Saratov
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - Yaroslavl Regional Hospital, Yaroslavl
- Spain (4):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital Univ. Central de Asturias, Oviedo
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
- Turkey (Türkiye) (7):
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Endokrinoloji, Adana
  - Aydın Adnan Menderes Üniversitesi Hastanesi, Aydin
  - Şişli Hamidiye Etfal Eğitim ve Araştırma Hastanesi- Seyrantepe Yerleşkesi- Endokrinoloji, Istanbul
  - Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi- Endokrinoloji, Istanbul
  - Haydarpaşa Numune Eğitim ve Araştırma Hastanesi - Endokrinoloji, Istanbul
  - Erciyes Üniversitesi Hastanesi- Nefroloji, Kayseri
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi - Kardiyoloji, Malatya
- United Kingdom (8):
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - Royal Derby Hospital, Derby
  - Western General Hospital, Edinburgh
  - Royal Surrey County Hospital - Diabetes, Guildford
  - Churchill Hospital, Oxford
  - Lister Hospital, Stevenage
  - Joint Clinical Research Facility - Swansea, Swansea

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Derived] Mohan V, Kesavadev J, Murthy LS, Anil G, Chandrappa M, Kar S, Mishra S. Efficacy and Safety of Once-Weekly Insulin Icodec in Indian Participants with Diabetes: Results from ONWARDS 1, 4, and 6 Studies. Diabetes Ther. 2025 Nov;16(11):2193-2212. doi: 10.1007/s13300-025-01799-4. Epub 2025 Oct 6. PMID 41051694
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Russell-Jones D, Babazono T, Cailleteau R, Engberg S, Irace C, Kjaersgaard MIS, Mathieu C, Rosenstock J, Woo V, Klonoff DC. Once-weekly insulin icodec versus once-daily insulin degludec as part of a basal-bolus regimen in individuals with type 1 diabetes (ONWARDS 6): a phase 3a, randomised, open-label, treat-to-target trial. Lancet. 2023 Nov 4;402(10413):1636-1647. doi: 10.1016/S0140-6736(23)02179-7. Epub 2023 Oct 17. PMID 37863084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 97 sites in 12 countries as follows (number of sites that screened subjects/ number of sites that randomized subject): Austria-(6/6), Canada-(5/5), Germany-(8/8), India-(6/6), Italy-(5/5), Japan-(7/7), Netherlands-(3/3), Russia-(10/10), Spain-(4/4), Turkey-(7/7), United Kingdom-(8/8), United States-(29/28).
Pre-assignment Details: This was a 52-week trial. The first 26 weeks of the trial constituted the main phase which was followed by a 26-week extension phase with focus on evaluating long term safety and provide long-term exposure data.
Groups:
- Insulin Icodec + Insulin Aspart: Participants received Insulin icodec along with Insulin aspart for 52 weeks subcutaneously. Participants received once weekly subcutaneous (s.c.) injection of Insulin icodec using PDS290 prefilled pen-injector at a starting dose of 7 times the pre-trial total daily basal insulin dose + 50% or 100% of their 7 times total daily basal insulin dose depending on insulin regime and HbA1c level. The following weekly dose was 7 times the total daily dose of the respective participants ('unit to unit switch' approach: current daily dose x 7). Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose reduced by 20 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 20 U. Dose titration of insulin aspart was based on the respective premeal(s) and bedtime self-measured plasma glucose (SMPG) measured weekly.
- Insulin Degludec + Insulin Aspart: Participants received Insulin degludec along with Insulin aspart for 52 weeks subcutaneously. Participants received once daily s.c. injection of Insulin degludec using PDS290 prefilled pen-injector at a dose in accordance with local label. Participants were to perform once daily SMPG. The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 millimoles per liter (mmol/L): dose reduced by 3 units (U); 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 3 U. Dose titration of insulin aspart was based on the respective premeal(s) and bedtime SMPG measured weekly.
Period: Main Phase (26 Weeks)
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Started | 290 | 292
Completed | 279 | 284
Not Completed | 11 | 8
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 9 | 7
Period: Extension Phase (26 Weeks)
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Started | 279 | 284
Completed | 274 | 281
Not Completed | 5 | 3
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart | Total
Number analyzed (Participants) | 290 | 292 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.08 (14.07) | 44.28 (14.07) | 44.18 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 120 | 245
  Male | 165 | 172 | 337
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 280 | 282 | 562
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 51 | 72 | 123
  Race: Black Or African American | 9 | 2 | 11
  Race: White | 230 | 218 | 448

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) at Week 26
Description: Change in HbA1c from baseline to week 26 is presented. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: Baseline (week 0), week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Percentage of HbA1c | -0.47 (0.07) | -0.51 (0.06)
Statistical Analysis 1: Comparison: Insulin Icodec + Insulin Aspart vs Insulin Degludec + Insulin Aspart; Change from baseline in HbA1c after 26 weeks was analysed using ANCOVA model with treatment, region, HbA1c group at screening and pre-trial basal insulin treatment as fixed factors, and baseline response as covariate; Test type: Non-Inferiority — Non-inferiority was considered confirmed if the estimated treatment difference was below 0.3%; p = 0.0065, ANCOVA; Treatment difference = 0.05, 95% CI 2-sided [-0.13 to 0.23]

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) at Week 52
Description: Change in HbA1c from baseline to week 52 is presented. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Percentage of HbA1c | -0.37 (0.05) | -0.54 (0.05)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline to week 26 is presented. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: Baseline (week 0), week 26
Population: Full analysis set included all randomised participants. Overall Number of Participants Analyzed = participants with available data.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/l)
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 276 | 287
millimoles per liter (mmol/l) | -0.84 (0.20) | -1.87 (0.20)

4. Secondary Outcome: Percentage of Time in Range 3.9-10.0 mmol/L (70-180 Milligrams Per Deciliter [mg/dL]) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time in range 3.9-10.0 mmol/L (70-180 mg/dL) using CGM system from week 22 to week 26 is presented. Time in range is defined as 100 times the number of recorded measurements in glycaemic range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive, divided by the total number of recorded measurements. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 261 | 272
Percentage of time | 59.10 (15.66) | 60.85 (15.03)

5. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQs) in Total Treatment Satisfaction
Description: Change in DTSQs in total treatment satisfaction from baseline to week 26 is presented. The sum score for DTSQ in total treatment satisfaction was calculated by adding the six item scores of items 1, 4, 5, 6, 7 and 8. The sum score for DTSQ can range from 0 to 36, with 0 being the lowest and 36 being the highest score in total treatment satisfaction. Higher scores on the DTSQ total score indicate higher treatment satisfaction. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: Baseline (week 0), week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 288 | 291
Score on a scale | 1.97 (0.27) | 3.06 (0.27)

6. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 26
Description: Number of severe hypoglycaemic episodes (level 3) from baseline to week 26 are presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Data is reported for 'main-on-treatment' period. The main-on-treatment period started at the date of first dose of trial product as recorded on the electronic case report form (eCRF), and ended at the first date of any of the following: the end date of the on-treatment period; week 26. On-treatment: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit, the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 26
Population: Safety analysis set included all participants who were randomly assigned to trial treatment and who took at least 1 dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 47 | 17

7. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 57
Description: Number of severe hypoglycaemic episodes (level 3) from baseline to week 57 are presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Data is reported for 'on-treatment' period. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 56 | 25

8. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL) Confirmed by Blood Glucose [BG] Meter): From Baseline (Week 0) to Week 26
Description: Number of clinically significant hypoglycaemic episodes (level 2) from baseline to week 26 are presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Data is reported for 'main-on-treatment' period. The main-on-treatment period started at the date of first dose of trial product as recorded on the eCRF, and ended at the first date of any of the following: the end date of the on-treatment period; week 26. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 2789 | 1478

9. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL) Confirmed by BG Meter): From Baseline (Week 0) to Week 57
Description: Number of clinically significant hypoglycaemic episodes (level 2) from baseline to week 57 are presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Data is reported for 'on-treatment' period. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 5047 | 2811

10. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 26
Description: Number of clinically significant hypoglycaemic episodes (level 2) or severe hypoglycaemic episodes (level 3) from baseline to week 26 presented. Clinically significant hypoglycaemia (level 2) is de-fined as plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypo-glycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring ex-ternal assistance for recovery. Data is reported for 'main-on-treatment' period, started at date of first dose of trial product as recorded on eCRF, and ended at first date of any of following: end date of on-treatment period; week 26. On-treatment period: Onset date on or after the first dose of trial product and no later than first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 2836 | 1495

11. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 57
Description: Number of clinically significant hypoglycaemic episodes (level 2) or severe hypoglycaemic episodes (level 3) from baseline to week 57 are presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Data is reported for 'on-treatment' period. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 5103 | 2836

12. Secondary Outcome: Number of Nocturnal Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 26
Description: Number of nocturnal clinically significant hypoglycaemic episodes (level 2) or severe hypogly-caemic episodes (level 3) from baseline to week 26 presented. Nocturnal: Period between 00:01 and 05:59 (both included). Clinically significant hypoglycaemia (level 2): Plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemia (level 3): Hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Data is reported for 'main-on-treatment' period, started at date of first dose of trial product as recorded on eCRF, and ended at first date of any of following: end date of on-treatment period; week 26. On-treatment period: Onset date on or after first dose of trial product and no later than first date of either fol-low-up visit, last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or end-date for in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 481 | 227

13. Secondary Outcome: Number of Nocturnal Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3): From Baseline (Week 0) to Week 57
Description: Number of nocturnal clinically significant hypoglycaemic episodes (level 2) or severe hypoglycaemic episodes (level 3) from baseline to week 57 are presented. Nocturnal: The period between 00:01 and 05:59 (both included). Clinically significant hypoglycaemia (level 2): Plasma glucose value of < 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemia (level 3): Hypoglycaemia with severe cognitive impairment requiring external assistance for recovery. Data is reported for 'on-treatment' period. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period. Data reflects total number of episodes across all participants within the arm.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 6
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
Episodes | 870 | 462

14. Secondary Outcome: Percentage of Time Spent Less Than (<) 3.0 mmol/L (54 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent < 3.0 mmol/L using CGM system from week 22 to week 26 is presented. Time spent below threshold (< 3.0 mmol/L [54 mg/dL]) was defined as 100 times the number of recorded measurements below the threshold, divided by the total number of recorded measurements. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 261 | 272
Percentage of time | 1.02 (1.64) | 0.68 (1.27)

15. Secondary Outcome: Percentage of Time Spent Greater Than (>) 10 mmol/L (180 mg/dL) Using Continuous Glucose Monitoring (CGM) System
Description: Percentage of time spent > 10 mmol/L using CGM system from week 22 to week 26 is presented. Time spent above threshold (> 10 mmol/L [180 mg/dL]) was defined as 100 times the number of recorded measurements above the threshold, divided by the total number of recorded measurements. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: From week 22 to week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 261 | 272
Percentage of time | 37.03 (16.21) | 36.25 (15.61)

16. Secondary Outcome: Mean Total Weekly Insulin Dose: From Week 24 to Week 26
Description: Mean total weekly insulin dose from week 24 to week 26 is presented. Data is reported for 'main-on-treatment' period. The main-on-treatment period started at the date of first dose of trial product as recorded on the eCRF, and ended at the first date of any of the following: the end date of the on-treatment period; week 26. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From week 24 to week 26
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 274 | 271
Units of insulin | 310.52 [295.70 to 326.08] | 322.68 [307.46 to 338.66]

17. Secondary Outcome: Mean Total Weekly Insulin Dose: From Week 50 to Week 52
Description: Mean total weekly insulin dose from week 50 to week 52 is presented. Data is reported for 'on-treatment' period. The on-treatment period: Onset date on or after the first dose of trial product and no later than the first date of either the follow-up visit (FU2), the last date on trial product + 5 weeks for once daily insulin and + 6 weeks for once weekly insulin or the end-date for the in-trial period.
Time Frame: From week 50 to week 52
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Units of insulin
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 273 | 269
Units of insulin | 310.14 [294.85 to 326.22] | 328.90 [312.86 to 345.75]

18. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 26 is presented. Data is reported for 'in-trial' period. In-trial observation period started at randomisation and ended at the date of: the last direct participant-site contact; withdrawal for participants who withdrew their informed consent; the last participant-investigator contact as defined by the investigator for participants who were lost to follow-up (i.e. possibly an unscheduled phone visit); death for participants who died before any of the above.
Time Frame: Baseline (week 0), week 26
Population: Full analysis set included all randomised participants.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
Number analyzed (Participants) | 290 | 292
kilograms | 1.29 (0.23) | 1.01 (0.23)

ADVERSE EVENTS:
Time Frame: Week 1 to week 57
Description: Treatment emergent adverse events (TEAEs) are reported: event that had onset date during on-treatment period: started 1st dose date of trial product as recorded on eCRF, and ended at 1st date of any of following: end of trial V56, last date on trial product+5 weeks for once daily insulin and+6 weeks for once weekly insulin, end-date for in-trial observation period. Safety analysis set: all participants randomly assigned to trial treatment who took at least 1 dose of trial product.
Arm/Group | Insulin Icodec + Insulin Aspart | Insulin Degludec + Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 1/290 | 0/292
Serious Adverse Events (participants affected / at risk) | 24/290 | 20/292
Other Adverse Events (participants affected / at risk) | 145/290 | 162/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec + Insulin Aspart (N=290) | Insulin Degludec + Insulin Aspart (N=292)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Brachiocephalic artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (13) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec + Insulin Aspart (N=290) | Insulin Degludec + Insulin Aspart (N=292)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 15 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 17 (31)
COVID-19 (Infections and infestations) | 74 (80) | 83 (88)
Diabetic retinopathy (Eye disorders) | 24 (28) | 26 (29)
Headache (Nervous system disorders) | 17 (27) | 16 (22)
Nasopharyngitis (Infections and infestations) | 48 (75) | 61 (84)
Pyrexia (General disorders) | 16 (22) | 20 (25)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT04848480/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT04848480/SAP_001.pdf